CLINICAL TRIAL: NCT03390790
Title: The Impact of Pre-procedure Periurethral Topical Lidocaine Application on Pain Scores After Complex Urodynamic Testing in Women
Brief Title: Lidocaine for Pain After Urodynamic Testing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, charbel salamon, Principal Investigator, Atlantic Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1112951-1
Record Dates: First submitted 2017-10-20; First posted 2018-01-04 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Voiding Disorders; Overactive Bladder; Urinary Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine gel (Experimental): If assigned to this arm, participants have lidocaine gel 2% applied to their external urethra and vagina one time prior to the urodynamics procedure.
  Interventions: Drug: Lidocaine gel 2%
- Lubricant gel (Placebo Comparator): If assigned to this arm, participants will have a standard lubricant gel applied to their external urethra and vagina prior to the urodynamics procedure.
  Interventions: Other: Standard lubricant gel

INTERVENTIONS:
Drug: Lidocaine gel 2% — If assigned to this intervention via randomization, participants will receive lidocaine (numbing) gel prior to their urodynamics procedure.
  Arms: Lidocaine gel
Other: Standard lubricant gel — If assigned to this intervention via randomization, participants will receive standard lubricant gel prior to their urodynamics procedure.
  Arms: Lubricant gel

SUMMARY:
Urodynamic testing can be associated with mild discomfort, particularly at the time of insertion, repositioning, and removal of the bladder catheter (a tube inserted into the bladder via the urethra). Few studies have investigated ways to improve patient comfort during this procedure. In this study, the investigators want to see if applying external lidocaine (a numbing gel) prior to the procedure can help to minimize patient discomfort.

DETAILED DESCRIPTION:
Urodynamic testing can be associated with mild discomfort, particularly at the time of insertion, repositioning, and removal of the bladder catheter (a tube inserted into the bladder via the urethra). Few studies have investigated ways to improve patient comfort during this procedure. In this study, the investigators want to see if applying lidocaine (a numbing gel) prior to the procedure can help to minimize patient discomfort.

Participation in this study will involve only 1 clinic visit (for urodynamic testing), plus 2 phone calls to ask participants about pain (1 at 4-6 hours after testing; and 1 at 24 hours after testing). Additionally, the investigators will record any adverse effects (such as an allergic reaction to the gel or new irritation/pain) that happen within 2 weeks after testing.

Participants will be randomly assigned to receive either lidocaine gel or placebo gel for their urodynamic testing. The placebo gel will be a standard lubricant gel, meaning that it contains no active drug. The assigned study regimen will be chosen by chance, like flipping a coin. Participants will have an equal (50/50) chance of being given either study regimen. Neither the participant nor the study doctor or nurse practitioner will know which study regimen the participant is getting. Additionally, a member of the study team will ask participants about their pain level before and after the testing. The rest of the urodynamic testing procedure will take place exactly as it would if the participant was not in this research study.

ELIGIBILITY:
Inclusion Criteria:

• All female patients between the ages of 40-80 undergoing urodynamic testing.

Exclusion Criteria:

* Urinary tract infection or symptoms of infection at time of procedure or within past 2 weeks
* History of urinary retention
* Known or suggested history of urethral syndrome or painful bladder syndrome
* Prior anti-incontinence surgery
* Prior pelvic surgery with placement of transvaginal mesh
* Known urethral or bladder anomaly including urethral diverticulum or congenital anomalies of the bladder or urethra
* History of genital herpes outbreak within the past 3 months
* Defects in mucosal surfaces including periurethral or vaginal abrasions, ulcerations, or lacerations
* Neurologic disease affecting urethral sensation
* Chronic pelvic pain
* Contraindication or allergy to topical anesthetic
* Pregnancy
* Syncopal episode during preparation for or execution of uroflowometry

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
The change in patient visual analog pain score (vaginal area only) from before procedure to 4-6 hours after urodynamic testing | Baseline and 4-6 hours post procedure.
  Participants will rate their pain according to a visual analog pain scale from 0 (no pain) to 100 (worst pain imaginable).

SECONDARY OUTCOMES:
Change in patient visual analog pain score (vaginal area only) from before procedure to 24 hours after urodynamic testing. | Baseline and 24 hours post procedure.
  Participants will rate their pain according to a visual analog pain scale from 0 (no pain) to 100 (worst pain imaginable).
Patient visual analog pain score (vaginal area only) before procedure, at conclusion of all procedure-related activities, 4-6 hours after procedure, and 24 hours after procedure. | Baseline and 24 hours post procedure.
  Participants will rate their pain according to a visual analog pain scale from 0 (no pain) to 100 (worst pain imaginable).
To assess voiding difficulties and other adverse events immediately after urodynamic testing, at 4-6 hours, 24 hours, and two weeks after urodynamic testing. | Baseline and 2 weeks post-procedure.
  Participants will receive a phone call at 4-6 hours and 24 hours after urodynamic testing. Any study participant-initiated complaints of voiding difficulties within two weeks of the procedure will be documented and addressed.
Urodynamic findings | At time of procedure.
  Standard urodynamics findings will be analyzed.
Procedure time | At time of procedure.
  Procedure time will be recorded for all subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantic Health System, Morristown, New Jersey, United States

REFERENCES:
- [Derived] Avondstondt AM, Chiu S, Salamon C. Periurethral Lidocaine Does Not Decrease Pain After Urodynamic Testing in Women: A Double-Blinded Randomized Control Trial. Female Pelvic Med Reconstr Surg. 2021 May 1;27(5):e528-e532. doi: 10.1097/SPV.0000000000000983. PMID 33208652